CLINICAL TRIAL: NCT05416047
Title: An Investigation of Frailty Markers and Outcomes in Patients Requiring Emergency Laparotomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Strathclyde (Other)
Responsible Party: Sponsor
Other Study IDs: GN20SG508
Record Dates: First submitted 2022-05-17; First posted 2022-06-13 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2022-06

CONDITIONS: Frailty; Surgery; Sarcopenia
MeSH Terms: conditions — Frailty; Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Frail and no frail: Frailty will be assessed using Rockwood Clinical Frailty Score
- Sarcopenia and no sarcopenia: Sarcopenia will be assessed using psoas muscle mass

SUMMARY:
Over 30,000 emergency abdominal operations (laparotomy, EmLAP) are performed in the UK annually and they are usually performed in adults over the age of 65. As such, it can be a risky operation with high chance of developing complications, including death, especially if there is frailty before the operation. Such patients are much more susceptible to infections or to have complications, such as wound breakdown, because of poor healing. Whilst some patients might be frail from the outset, surgery can cause patients to become frail ('surgical frailty'). This can happen in all age groups, not just the elderly and is not uncommon after an EmLap.

This study aims to establish blood tests (biomarkers) associated with frailty, explore the ability of frailty markers measured before EmLAP to predict death after EmLAP, define changes in frailty in EmLAP patients and analyse the influence of frailty on quality of life post EmLAP.

Over 2 years, 150 patients age ≥40 undergoing EmLAP in a hospital will be recruited and followed up for 90 days looking at different frailty markers. These include (a)blood tests (biomarkers) analysed in a special laboratory machine called mass spectrometer to identify chemical markers linked to frailty status (b)CT scan looking at muscle bulk (sarcopenia) (c)Rockwood Clinical Frailty Score, a scoring system assessing how much a patient can do (1 is fit; 9 is extremely frail).

The investigators hope that these results will improve our understanding of frailty and lead to further research to improve outcomes for EmLAP patients.

DETAILED DESCRIPTION:
Over 30,000 emergency laparotomies (EmLAP) are performed in the UK annually yet research in EmLAP is sparse. The largest UK national observational cohort study (Emergency Laparotomy and frailty study, ELF) found higher rates of 30 and 90-day mortality as well as higher post-operative complications in the frail patients. These findings were reflected in the National Emergency Laparotomy Audit (NELA) 7th report and the results have worsened.

Frailty is a clinical syndrome of increased vulnerability that results from ageing associated multi-system physiological decline resulting in reduction of the individual's ability to cope with physiological stress such as surgery. Frailty can be identified using different assessments but due to practicality in emergency setting, the Rockwood Clinical Frailty Score (CFS) is increasingly used and has been incorporated in NELA. Frailty is not unique to the older EmLAP population, it is also present in 16% of adults aged 40 to 65 years. If frailty pre-EmLAP is prevalent, then it must be remembered that surgery can induce frailty in non-frail patients and worsening frailty in those that were already frail (surgical frailty).

Overall, there is lack of understanding in the biochemical aetiology of frailty. Early detection of subclinical changes and changes at the molecular level are key to enhancing our understanding of the biology of frailty and ultimately improving patients outcomes. This study aims to establish blood based biomarkers that could identify frailty objectively in EmLAP patients. The secondary aims are to compare preoperative frailty markers in their ability to predict 30 and 90-day mortality post-EmLAP, define perioperative changes in frailty in patients undergoing EmLAP and analyse the influence of perioperative frailty on morbidity and quality of life post- EmLAP.

Methods A prospective single centred observational study will be conducted over on 150 patients ≥40 years of age that undergo EmLAP over 2years. Patients will be included according to the established NELA criteria. The variables collected include demographics, co-morbidities using, polypharmacy, lifestyle, place of residence, indication and type of surgery (as per NELA criteria) and prognostic NELA score.

The frailty markers will be collected preoperatively and post- operatively day 1 and 7:

1. Blood sample for mass spectrometry analysis (additional blood tube on top of routine bloods)
2. Preoperative CT abdomen pelvis
3. Malnutrition Universal Screening Tool (MUST) score (recorded on admission)
4. Abbreviated Mental Test (AMT) score (recorded on admission)
5. Routine serum biochemistry and haematology: Hb, White cells, C- Reactive protein, Albumin
6. Rockwood Clinical Frailty Score (CFS). Score 1 -9 with frail as ≥4.

Other follow-up data collection:

1. Day 30 and 90 mortality assessed from medical records
2. Place of residence post discharge following EmLAP
3. Day 30 and 90 blood samples for mass spectrometry analysis
4. 30 day morbidity (according Clavien Dindo classification)
5. Total hospital stay including critical care stay
6. Day 30 and 90 quality of life post EmLAP using EQ5D-5L.

The frailty markers will be compared between groups of frail and non-frail patients using statistical methods such as regression model and adjust for appropriate confounding variables.

ELIGIBILITY:
Inclusion Criteria:

* Over 40 years of age
* NELA/ ELLSA inclusion criteria:
* Open, laparoscopic, or laparoscopically-assisted procedures
* Procedures involving the stomach, small or large bowel, or rectum for conditions such as perforation, ischaemia, abdominal abscess, bleeding or obstruction
* Washout/evacuation of intra-peritoneal abscess (unless due to appendicitis or cholecystitis - excluded, see below)
* Washout/evacuation of intra-peritoneal haematoma
* Bowel resection/repair due to incarcerated incisional, umbilical, inguinal and femoral hernias (but not hernia repair without bowel resection/repair). E.g. Large incisional hernia repair with bowel resection Bowel resection/repair due to obstructing/ incarcerated incisional hernias provided the presentation and findings were acute. This will include large incisional hernia repair with division of adhesions.
* Laparotomy/laparoscopy with inoperable pathology (e.g. peritoneal/hepatic metastases) where the intention was to perform a definitive procedure. This does not include purely diagnostic procedures.
* Laparoscopic/Open Adhesiolysis
* Return to theatre for repair of substantial dehiscence of major abdominal wound (i.e. "burst abdomen")
* Any reoperation/return to theatre for complications of elective general/upper GI surgery meeting the criteria above is included. Returns to theatre for complications following non-GI surgery are now excluded (see exclusion criteria below).

Exclusion Criteria:

* Under 40 years of age
* CT scan or postoperative finding of inoperable disseminated peritoneal disease
* Open and close laparotomy (postoperative palliation, non-survivable global ischemia where there are <90cm from duodenojejunal junction to stoma)
* Complication from colonic stenting requiring laparotomy
* NELA exclusion criteria:
* Elective laparotomy / laparoscopy
* Diagnostic laparotomy/laparoscopy where no subsequent procedure is performed (NB, if no procedure is performed because of inoperable pathology, then include)
* Appendicectomy +/- drainage of localised collection unless the procedure is incidental to a non-elective procedure on the GI tract
* Cholecystectomy +/- drainage of localised collection unless the procedure is incidental to a non-elective procedure on the GI tract (All surgery involving the appendix or gallbladder, including any surgery relating to complications such as abscess or bile leak is excluded. The only exception to this is if carried out as an incidental procedure to a more major procedure. There might be extreme cases of peritoneal contamination, but total exclusion avoids subjective judgement calls about severity of contamination.)
* Non-elective hernia repair without bowel resection or division of adhesions
* Minor abdominal wound dehiscence unless this causes bowel complications requiring resection.
* Non-elective formation of a colostomy or ileostomy as either a trephine or a laparoscopic procedure (NB: if a midline laparotomy is performed, with the primary procedure being formation of a stoma then this should be included)
* Vascular surgery, including abdominal aortic aneurysm repair
* Caesarean section or obstetric laparotomies
* Gynaecological laparotomy
* Ruptured ectopic pregnancy, or pelvic abscesses due to pelvic inflammatory disease
* Laparotomy/laparoscopy for pathology caused by blunt or penetrating trauma
* All surgery relating to organ transplantation (including returns to theatre for any reason following transplant surgery)
* Surgery relating to sclerosing peritonitis
* Surgery for removal of dialysis catheters
* Laparotomy/laparoscopy for oesophageal pathology
* Laparotomy/laparoscopy for pathology of the spleen, renal tract, kidneys, liver, gall bladder and biliary tree, pancreas or urinary tract
* Returns to theatre for complications (eg bowel injury, haematoma, collection) following non-GI surgery are now excluded. i.e returns to theatre following renal, urological, gynaecological, vascular, hepatic, pancreatic, splenic surgery are excluded

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing emergency laparotomy in Royal Alexandra Hospital
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-05-30 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Preoperative frailty markers | 30 days
  Recruited patients will be categorised into frail and non- frail group according to collected data on co-morbidities, CT measurement for sarcopenia, Rockwood CFS and frailty questionnaires results. Biomarker identified on mass spectrometry will be compared with result from patient grouping of frail and non- frail.

SECONDARY OUTCOMES:
Perioperative changes on 30- day morbidity, 30-day and 90-day mortality | 90 days
  Data on length of total hospital stay, length of stay in critical care, post operative complications according to Clavien Dindo Classification, time from surgery to medical discharge (i.e. when medically well, excluding social issues etc), date and cause of death within 90 days post operative will be collected and compared among frail and non- frail group of patients.
Influence of perioperative frailty on quality of life post emergency laparotomy | 90 days
  Changes in quality of life post EmLAP and place of residence post discharge will be explored using EQ5D-5L questionnaire on day 30 and 90 post operative

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Alexandra Hospital, Paisley, Renfrewshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ng HJ, Rattray NJW, Quasim T, Moug SJ. Changes in frailty status and discharge destination post emergency laparotomy. World J Emerg Surg. 2025 Apr 25;20(1):37. doi: 10.1186/s13017-025-00612-8. PMID 40281633
- [Derived] Ng HJ, Quasim T, Rattray NJW, Moug S. Investigation of frailty markers including a novel biomarker panel in emergency laparotomy: protocol of a prospective cohort study. BMC Surg. 2023 Jul 5;23(1):190. doi: 10.1186/s12893-023-02093-5. PMID 37408022